CLINICAL TRIAL: NCT05311579
Title: Efficacy and Safety of Niraparib in Combination With Anlotinib Based on CA 125 Level in Newly Diagnosed Ovarian Cancer: A Open-label, Single Arm, Prospective Phase II Trial
Brief Title: Niraparib Plus Anlotinib for Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIRAN1
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Ovarian Carcinoma; Survival Outcomes; Adverse Events; Niraparib; Anlotinib; CA125; Chemotherapy; Targeted Therapy; Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian cancer patients with increased CA125 (Experimental): Patients with CA125 >35 U/ml or increased to 2 x nadir, and with no evidence of imaging recurrence after completion of 1st-line platinum-based chemotherapy
  Interventions: Combination Product: Niraparib plus anlotinib

INTERVENTIONS:
Combination Product: Niraparib plus anlotinib — Niraparib QD D1-21 plus Anlotinib 10mg QD D1-14 until disease progression or intolerable toxicity
  21days/cycle

SUMMARY:
This is a phase II trial to explore efficacy and safety of niraparib in combination with anlotinib based on CA 125 level in newly diagnosed ovarian cancer. After completion of 1st-line platinum-based chemotherapy with a normal CA-125 concentration, in patients with CA-125 increased > 35U/ml, and with no evidence of imaging recurrence, niraparib and anlotinib are used as 1st maintenance therapy for newly diagnosed advanced ovarian cancer after achieving complete or partial remission to platinum-containing chemotherapy. The primary objective of this study is to explore the efficacy of niraparib combined with anlotinib based on CA 125 level in newly diagnosed ovarian cancer with no evidence of imaging recurrence. A total o f36 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion criteria

1. Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent
2. Patients must be female ≥18 years of age
3. Patients must have histologically diagnosed non-mucinous ovarian cancer that is Stage III or IV according to FIGO criteria, and niraparib is used as 1st maintenance therapy after achieving CR/PR to front-line platinum-containing chemotherapy
4. After completion of front-line platinum-based chemotherapy with a normal CA-125 concentration: CA-125 increased > 35U/ml on 2 occasions (Repeat CA 125 any time but normally not less than 1 week after the first elevated CA 125 level), and with no evidence of imaging recurrence
5. After completion of front-line platinum-based chemotherapy, CA125 decreased by 90% and was not in the normal range: the level of CA125 at the end of chemotherapy as the nadir, CA-125 increased to 2 x nadir on 2 occasions (Repeat CA 125 any time but normally not less than 1 week after the first elevated CA 125 level), and with no evidence of imaging recurrence
6. Allow to combinate bevacizumab during front-line chemotherapy
7. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Patients must have adequate organ function, defined as follows:

   * Absolute neutrophil count ≥ 1,500/μL
   * Platelets ≥ 100,000/μL
   * Hemoglobin ≥ 10 g/dL
   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault equation
   * Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ 1 x ULN
   * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
9. Pregnancy test results were negative and patients willing to use appropriate contraceptive methods while in the trial and within 3 months after the last dose of this study treatment; or keep abstinence during the trial; or women with no potential fertility.
10. Ability to comply with protocol.
11. All of the adverse events caused by chemotherapy recovered to Common Terminology Criteria Adverse Events (CTCAE) grade 1 or baseline, except for stable sensory neuropathy or hair loss ≤ CTCAE grade 2.

Exclusion criteria

1. Allergy to active or inactive ingredients of niraparib or drugs with similar chemical structures.
2. Allergy to active or inactive ingredients of anlotinib or drugs with similar chemical structures.
3. Active and uncontrollable brain metastasis or leptomeningeal metastasis. Patients with spinal cord compression can still be considered if they have received targeted treatment and have evidence of clinical stability of the disease for at least > 28 days (controlled brain metastasis must have received radiotherapy or chemotherapy at least 1 month prior to study entry; patients may not have new symptoms related to brain lesions or symptoms indicating disease progression and either take stable dose of hormone or do not need to take hormone).
4. Major surgery performed within 3 weeks before enrollment, or any surgical effects that have not recovered from the surgery, or chemotherapy.
5. Palliative radiotherapy encompassing >20% of the bone marrow within 1 week of the first dose of study treatment
6. Any other malignant tumor exclude ovarian cancer has been diagnosed within 2 years before enrollment (except for completely treated basal or squamous cell skin cancer).
7. Current or previous myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
8. Other severe or uncontrolled diseases, including but not limited to:

   * Uncontrollable nausea and vomiting, inability to swallow study drug, and any gastrointestinal disease that may interfere with the absorption and metabolism of the drug
   * Active viral infections, such as human immunodeficiency virus, hepatitis B virus, hepatitis C virus and so on
   * Uncontrolled epileptic seizures, unstable spinal cord compression, superior vena cava syndrome or other psychiatric disorders that may affect patients' informed consent
   * Immunodeficiency (except for splenectomy), or other diseases that investigators believe may expose patients to high-risk toxicity.
9. Have the risk or tendency of bleeding and history of thrombosis

   * CTCAE grade 2 bleeding event occurred within 3 months prior to screening or CTCAE ≥ grade 3 bleeding event occurred within 3 months prior to screening
   * Have history of gastrointestinal bleeding or confirmed bleeding tendency within 6 months prior to screening. e.g. esophageal varices with bleeding risk, local active ulcer focus or fecal occult blood above ++
   * Have active bleeding or coagulation dysfunction, have bleeding risk or undergoing thrombolytic or anticoagulant therapy
   * Need anticoagulant therapy with warfarin or heparin
   * Need long-term anti-platelet therapy (e.g. aspirin, clopidogrel)
   * Have occurred thrombus or embolism event in past 6 months, e.g. cerebral vascular accident（including transient cerebral ischemic attack), pulmonary embolism
10. A history of severe cardiovascular disease:

    * New York Heart Association (NYHA) grade 3/4 congestive heart failure (CHF)
    * Unstable angina or newly diagnosed angina/myocardial infarction within 12 months prior to screening
    * Cardiac arrhythmia despite need medication (patients taking β-receptor blockers or digoxin can be enrolled)
    * CTCAE ≥ grade 2 valvular heart disease
    * Poorly controlled hypertension (systolic pressure>150 mmHg or diastolic pressure>100 mmHg)
11. The following laboratory indexed are abnormal:

    * Hyponatremia (serum sodium < 130 mmol/L); baseline serum potassium < 3.5 mmol/L (potassium supplements can be used to restore serum potassium above this before enrollment)
    * Thyroid dysfunction and cannot maintain normal despite medical treatment
12. Previous/current diseases and treatment or abnormal laboratory indexed those interfere with study result or participation of the whole study; or the investigator confirmed not suitable for this trial; have platelet or red blood cell transfusion within 4 weeks prior to the first dose of study treatment
13. Patients must not be pregnant, breastfeeding, or expecting to conceive children, while receiving study treatment
14. Corrected QT interval（QTc>450 milliseconds); if patients have QTc prolongation because of cardiac pacemaker confirmed by investigator and no other cardiac disorder, whether enrollment need further discussion with investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-03-27 (Estimated); Study Completion 2024-03-27 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 24 months
  Progression free survival (PFS) by RECIST v 1.1

SECONDARY OUTCOMES:
Time to first subsequent therapy (TFST) | 24 months
  Time to first subsequent therapy (TFST)
Overall survival (OS) | 48 months
  Overall survival (OS)
Adverse events | 24 months
  Adverse event (AE), Treatment emergent adverse event (TEAE), Serious adverse event (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China